CLINICAL TRIAL: NCT00084422
Title: A Phase I Study Of CEP-701 In Patients With Refractory Neuroblastoma (IND # 67,722)
Brief Title: N2001-03: CEP-701 in Treating Young Patients With Recurrent or Refractory High-Risk Neuroblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: New Approaches to Neuroblastoma Therapy Consortium (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000363630; P01CA081403 (NIH); NANT-2001-03
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Neuroblastoma
Keywords: recurrent neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — lestaurtinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Group (Experimental)
  Interventions: Drug: lestaurtinib

INTERVENTIONS:
Drug: lestaurtinib — Given orally twice daily x 5 consecutive days followed by a two day rest. 28 days = 1 treatment course. Courses repeated indefinitely without gap provided patient has recovered course from toxicities and no DLTs. Dose level assigned according to the planned dose escalation schedule.
  Other Names: CEP-701

SUMMARY:
RATIONALE: CEP-701 may stop the growth of tumor cells by blocking the enzymes necessary for their growth.

PURPOSE: This phase I trial is studying the side effects and best dose of CEP-701 in treating young patients with recurrent or refractory high-risk neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of CEP-701 in pediatric patients with recurrent or refractory high-risk neuroblastoma.
* Determine the dose-limiting toxicity of this drug in these patients.
* Determine the pharmacokinetic behavior of this drug in these patients.

Secondary

* Determine the degree of TrkB tyrosine kinase inhibition activity present in the serum of patients treated with this drug.
* Correlate the degree of TrkB tyrosine kinase inhibition activity in these patients with dose level, pharmacokinetics, and antitumor activity data of this drug.
* Determine the antitumor activity of this drug in these patients.

OUTLINE: This is an open-label, dose-escalation, multicenter study.

Patients receive oral CEP-701 twice daily* on days 1-5, 8-12, 15-19, and 22-26. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

NOTE: *On day 1 of course 1 only, patients receive oral CEP-701 once instead of twice.

Cohorts of 3-6 patients receive escalating doses of CEP-701 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, the dose level is expanded up to 9 patients.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of neuroblastoma confirmed by at least 1 of the following:

  * Histology
  * Demonstrates clumps of tumor cells in the bone marrow with elevated urinary catecholamine metabolites
* Recurrent or resistant/refractory disease
* Neuroblastoma metastatic to the bone marrow with granulocytopenia, anemia, and/or thrombocytopenia allowed
* High-risk disease
* Patients in first response after completion of a prior front-line myeloablative regimen OR who were medically ineligible to receive a front-line myeloablative regimen must meet at least 1 of the following criteria:

  * Viable neuroblastoma determined by biopsy of a persistent lesion as seen on CT scan, MRI, or metaiodobenzylguanidine (MIBG) scan

    * If lesion was irradiated, biopsy must be performed at least 4 weeks after completion of prior radiotherapy
  * Morphologic evidence of tumor in bone marrow
* Second or greater response (without histologic confirmation) allowed
* Meets at least 1 of the following criteria:

  * At least 1 unidimensionally measurable lesion on CT scan, MRI, or X-ray

    * At least 20 mm by conventional techniques OR at least 10 mm by spiral CT scan
  * MIBG scan with positive uptake at a minimum of 1 site
  * Bone marrow with tumor cells on routine morphology (not by NSE staining only) of bilateral aspirate and/or biopsy AND/OR at least 5 tumor cells/10^6 mononuclear cells in the bone marrow by immunocytologic analysis of 2 consecutive bone marrows performed at least 1 day but no more than 4 weeks apart

PATIENT CHARACTERISTICS:

Age

* 21 and under at diagnosis

Performance status

* Karnofsky 50-100% (for patients > 16 years of age)
* Lansky 50-100% (for patients ≤ 16 years of age)

Life expectancy

* More than 2 months

Hematopoietic

* See Disease Characteristics
* Absolute neutrophil count ≥ 1,000/mm^3
* Platelet count ≥ 50,000/mm^3 (transfusion independent)
* Hemoglobin ≥ 8.0 g/dL (red blood cell transfusions allowed)

Hepatic

* ALT and AST ≤ 3.0 times upper limit of normal (ULN)
* Total bilirubin ≤ 1.5 times ULN

Renal

* Creatinine ≤ 1.5 times normal OR
* Creatinine clearance or radioisotope glomerular filtration rate ≥ 60 mL/min

Cardiovascular

* Ejection fraction ≥ 50% by echocardiogram or MUGA OR
* Fractional shortening ≥ 28% or above lower limit of normal by echocardiogram

Pulmonary

* Lung function normal
* No dyspnea at rest
* No exercise intolerance
* No supplemental oxygen requirement

Other

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception
* No uncontrolled infection
* No other concurrent illness that would preclude study treatment

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Chemotherapy
* At least 2 weeks since prior biologic or non-myelosuppressive therapy and recovered
* More than 7 days since prior growth factors
* No prior allogeneic stem cell transplantation AND no extensive chronic graft-versus-host disease
* No concurrent growth factors except filgrastim (G-CSF) or sargramostim (GM-CSF) administered for neutropenia lasting for more than 7 days or for confirmed or clinical septicemia associated with neutropenia

Chemotherapy

* At least 3 months since prior myeloablative chemotherapy with stem cell transplantation
* At least 2 weeks since prior chemotherapy and recovered

Endocrine therapy

* No concurrent corticosteroid therapy except replacement therapy for adrenal insufficiency or treatment for increased intracranial pressure

Radiotherapy

* See Disease Characteristics
* Recovered from prior radiotherapy
* At least 6 weeks since prior therapeutic-dose MIBG
* At least 6 weeks since prior craniospinal or other radiotherapy involving significant bone marrow (i.e., total pelvis or total abdomen)
* At least 4 weeks since prior radiotherapy to any site biopsied
* At least 2 weeks since prior local palliative radiotherapy (small port)

Surgery

* Not specified

Other

* No prior CEP-701
* No concurrent administration of any of the following CYP3A4 inhibitors:

  * Cyclosporine
  * Clotrimazole
  * Ketoconazole
  * Erythromycin
  * Clarithromycin
  * Troleandomycin
  * HIV protease inhibitors
  * Nefazodone
  * Itraconazole
  * Voriconazole

Ages: 1 Day to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 47 (Actual)
Dates: Start 2003-08; Primary Completion 2009-09 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) of CEP-701 given on a twice daily chronic administration schedule (two days on , two days off) to children with high risk relapsed or residual neuroblastoma. | Within 28 days of treatment at each dose level.
To determine dose limiting toxicities (DLTs) of CEP-701 given on this schedule | Within first 28 days of therapy.
To characterize the pharmacokinetic (PK) behavior of CEP-701 in children with residual or refractory high-risk neuroblastoma. | Days 1,5 and 26 of first course only.
  Participation in PK studies is voluntary and not a requirement for study entry.

SECONDARY OUTCOMES:
To determine the degree of TrkB tyrosine kinase inhibition activity present in the serum of patients treated with CEP-701, and correlate these findings with dose level, pharmacokinetic and anti-tumor activity data. | Days 1,5 and 26 of first course only.
To define the antitumor activity of CEP-701, within the confines of a Phase I study. | Evaluation at end of courses 1, 2, 4 and then every 4 courses until patient goes off therapy.

CONTACTS AND LOCATIONS:
Overall Officials: John M. Maris, MD, Principal Investigator — Children's Hospital of Philadelphia; Garrett M. Brodeur, MD, Study Chair — Children's Hospital of Philadelphia
Locations (12):
- United States (11):
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Lucille Salter Packer Children's Hospital, Stanford University, Palo Alto, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - AFLAC Cancer Center and Blood Disorders Service of Children's Healthcare of Atlanta - Egleston Campus, Atlanta, Georgia
  - University of Chicago Comer Children's Hospital, Chicago, Illinois
  - Children's Hospital Boston, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Morgan Stanley Children's Hospital of New York-Presbyterian, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
- Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Result] Minturn JE, Villablanca J, Yanik GA, et al.: Phase I trial of lestaurtinib for children with refractory neuroblastoma (NB): A New Approach to Neuroblastoma Therapy (NANT) Consortium study. [Abstract] J Clin Oncol 28 (Suppl 15): A-9532, 2010.
- [Result] Maris J, Minturn J, Evans A, et al.: Phase I trial of the orally bioavailable TRK tyrosine kinase inhibitor CEP-701 in refractory neuroblastoma: a New Approaches to Neuroblastoma Therapy (NANT) study. [Abstract] Pediatr Blood Cancer 45 (4 Suppl 1): A-0.129, 416, 2005.